CLINICAL TRIAL: NCT01993836
Title: Markers of Alzheimers Disease and Cognitive Outcomes After Perioperative Care
Acronym: MADCO-PC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00045180
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Alzheimers Disease; Postoperative Delirium; Post Operative Cognitive Dysfunction
Keywords: isoflurane; propofol; total intravenous anesthesia; inhaled anesthetic; volatile anesthetic; anesthesia; delirium; Post Operative Cognitive Dysfunction; Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Emergence Delirium; Delirium; Cognitive Dysfunction | interventions — Propofol; Anesthesia, General; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Intravenous Anesthesia with Propofol (Active Comparator): Patients in this arm will receive general anesthesia with propofol as the primary amnestic agent.
  Interventions: Drug: Total intravenous anesthesia with propofol
- General anesthesia with Isoflurane (Active Comparator): Patients in this arm will undergo general anesthesia with isoflurane as the primary amnestic agent.
  Interventions: Drug: General anesthesia with isoflurane

INTERVENTIONS:
Drug: Total intravenous anesthesia with propofol
  Arms: Total Intravenous Anesthesia with Propofol
Drug: General anesthesia with isoflurane
  Arms: General anesthesia with Isoflurane

SUMMARY:
This study will examine the hypothesis that changes in the cognition (i.e. thinking and memory) after anesthesia and surgery are correlated with changes in markers of Alzheimers Disease in the fluid around the brain and spinal cord (i.e. cerebrospinal fluid, or CSF), and/or changes in brain connectivity. The investigators will also examine whether different types of anesthesia have different effects on these CSF markers of Alzheimers disease, or different effects on thinking and memory after anesthesia and surgery, or differential effects on the correlation between cognitive changes and CSF marker changes.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients 60 years of age or older
* Surgery scheduled to last at least 2 hours (including time for anesthesia induction, etc)
* English speaking ability.
* Ability to give informed consent

Exclusion Criteria:

* Inmate of a correctional facility (i.e. prisoners).
* Pregnancy
* Documented or suspected family or personal history of malignant hyperthermia.
* Patient unable to receive either propofol or isoflurane due to allergy or other specific contraindication.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, PhD, Principal Investigator — Duke University Medical Center, Anesthesiology Department, Neuroanesthesia Division
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Villalobos D, Reese M, Wright MC, Wong M, Syed A, Park J, Hall A, Browndyke JN, Martucci KT, Devinney MJ, Acker L, Moretti EW, Talbot L, Colin B, Ohlendorf B, Waligorska T, Shaw LM, Whitson HE, Cohen HJ, Mathew JP, Berger M. Perioperative changes in neurocognitive and Alzheimer's disease-related cerebrospinal fluid biomarkers in older patients randomised to isoflurane or propofol for anaesthetic maintenance. Br J Anaesth. 2023 Aug;131(2):328-337. doi: 10.1016/j.bja.2023.04.019. Epub 2023 Jun 2. PMID 37271721
- [Derived] Berger M, Browndyke JN, Cooter Wright M, Nobuhara C, Reese M, Acker L, Bullock WM, Colin BJ, Devinney MJ, Moretti EW, Moul JW, Ohlendorf B, Laskowitz DT, Waligorska T, Shaw LM, Whitson HE, Cohen HJ, Mathew JP; MADCO-PC Investigators. Postoperative changes in cognition and cerebrospinal fluid neurodegenerative disease biomarkers. Ann Clin Transl Neurol. 2022 Feb;9(2):155-170. doi: 10.1002/acn3.51499. Epub 2022 Feb 1. PMID 35104057

RESULTS

PARTICIPANT FLOW:
Groups:
- General Anesthesia With Isoflurane: Surgical patients randomized to receive inhalational anesthesia with isoflurane during surgery
- Total Intravenous Anesthesia With Propofol: Surgical patients randomized to receive intravenous anesthesia with propofol during surgery
- Non-Surgical Controls: Cohort of community dwelling healthy controls for tertiary comparison
Period: Overall Study
Arm/Group | General Anesthesia With Isoflurane | Total Intravenous Anesthesia With Propofol | Non-Surgical Controls
Started | 72 (This represents the number of enrolled patients who completed baseline cognitive testing) | 68 | 51
Completed | 55 | 55 | 46
Not Completed | 17 | 13 | 5
Not completed — Surgery Cancelled | 3 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Withdrawal by Subject | 12 | 10 | 5

BASELINE CHARACTERISTICS:
Population: Subjects who returned for six-week follow-up visit.
Groups:
- Total Intravenous Anesthesia With Propofol: Surgical patients randomized to receive iintravenous anesthesia with propofol during surgery
- Total: Total of all reporting groups
Arm/Group | General Anesthesia With Isoflurane | Total Intravenous Anesthesia With Propofol | Non-Surgical Controls | Total
Number analyzed (Participants) | 55 | 55 | 46 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (6.1) | 69.7 (6.9) | 69.6 (7.6) | 69.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 18 | 59
  Male | 38 | 31 | 28 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 8 | 9 | 19
  White | 52 | 47 | 36 | 135
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 46 | 156
Baseline CSF levels [Median (Full Range); unit: pg/ml]
  Tau | 47 [24 to 108] | 50 [23 to 108] | 58.5 [34 to 88] | 49 [23 to 108]
  Abeta | 369 [140 to 466] | 352 [178 to 472] | 330.5 [169 to 592] | 347 [140 to 592]
  P-Tau | 26 [10 to 52] | 28 [11 to 52] | 21.0 [16 to 29] | 25 [10 to 52]
Baseline CSF ratio levels [Median (Full Range); unit: ratio]
  Tau/Abeta Ratio | 0.13 [0.06 to 0.69] | 0.14 [0.06 to 0.55] | 0.16 [0.11 to 0.28] | 0.14 [0.06 to 0.69]
  P-Tau/Abeta Ratio | 0.08 [0.03 to 0.27] | 0.08 [0.03 to 0.25] | 0.06 [0.04 to 0.10] | 0.07 [0.03 to 0.27]

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Perioperative Change in Cerebrospinal Fluid (CSF) Markers of Alzheimers Disease and Perioperative Cognitive Change
Description: Spearman correlation was used here as the CSF markers follow a skewed distribution. Spearman correlation describes the strength of the monotonic relationship between two measures and is bounded between -1 and 1. Negative values indicate an inverse relationship while positive values mean that the variables move in tandem.
Time Frame: Baseline to 6 weeks
Population: Analysis for the primary and secondary outcome 6 use the combination of both randomized treatment groups. The treatment groups are separated and compared in secondary analysis of outcomes 3-5, and the control group is only used in tertiary analyses. To be included in the outcome analysis patients must have returned for six-week follow-up visit.
Measure: Median (Full Range); unit: pg/ml
Groups:
- Combined Surgical Cohort: The combination of both surgical randomized treatment groups.
Arm/Group | Combined Surgical Cohort
Number analyzed (Participants) | 110
pg/ml
  Tau | -1.21 [-26 to 32]
  Abeta | -5.09 [-189 to 211]
  P-Tau | -0.44 [-31 to 85]
Statistical Analysis 1: Comparison: Combined Surgical Cohort; Correlation between 6-week change in Tau and continuous cognitive index; Test type: Other; Spearman Correlation = -0.03, 95% CI 2-sided [-0.23 to 0.18]
Statistical Analysis 2: Comparison: Combined Surgical Cohort; Correlation between 6-week change in Abeta and continuous cognitive index; Test type: Other; Spearman Correlation = -0.08, 95% CI 2-sided [-0.29 to 0.13]
Statistical Analysis 3: Comparison: Combined Surgical Cohort; Correlation between 6-week change in P-Tau and continuous cognitive index; Test type: Other; Spearman Correlation = 0.12, 95% CI 2-sided [-0.08 to 0.32]

2. Primary Outcome: Correlation Between Perioperative Change in Ratios of Cerebrospinal Fluid (CSF) Markers of Alzheimers Disease and Perioperative Cognitive Change
Description: Spearman correlation was used here as the ratio of CSF markers follow a skewed distribution. Spearman correlation describes the strength of the monotonic relationship between two measures and is bounded between -1 and 1. Negative values indicate an inverse relationship while positive values mean that the variables move in tandem.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: ratio
Arm/Group | Combined Surgical Cohort
Number analyzed (Participants) | 110
ratio
  Tau/Abeta Ratio | 0.001 [-0.20 to 0.21]
  P-Tau/Abeta Ratio | 0.002 [-0.10 to 0.41]
Statistical Analysis 1: Comparison: Combined Surgical Cohort; Correlation between 6-week change in Tau/Abeta ratio and continuous cognitive index; Test type: Other; Spearman Correlation = 0.02, 95% CI 2-sided [-0.19 to 0.22]
Statistical Analysis 2: Comparison: Combined Surgical Cohort; Correlation between 6-week change in P-Tau/Abeta ratio and continuous cognitive index; Test type: Other; Spearman Correlation = 0.16, 95% CI 2-sided [-0.05 to 0.34]

3. Secondary Outcome: Continuous Cognitive Index Score Change Difference Between Anesthetic Agent Groups
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a factor analysis was performed on the 10 cognitive test scores from baseline. To quantify overall cognitive function, a baseline cognitive index was first calculated as the mean of the preoperative domain scores. The cognitive index score has a mean of zero, thus any positive score is above the mean, any negative score is below the mean. A continuous change score was then calculated by subtracting the baseline from the 6-week cognitive index. A negative change score indicating decline and a positive score indicating improvement. The resulting outcome measure is unbounded with a standard deviation of 0.31 in the full surgical cohort.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Total Intravenous Anesthesia With Propofol: Patients in this arm will receive general anesthesia with propofol as the primary amnestic agent.
  Total intravenous anesthesia with propofol
- General Anesthesia With Isoflurane: Patients in this arm will undergo general anesthesia with isoflurane as the primary amnestic agent.
  General anesthesia with isoflurane
Arm/Group | Total Intravenous Anesthesia With Propofol | General Anesthesia With Isoflurane
Number analyzed (Participants) | 55 | 55
units on a scale | 0.019 (0.05) | 0.061 (0.04)
Statistical Analysis 1: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Test type: Other; p = 0.360, t-test, 2 sided

4. Secondary Outcome: Change in CSF Markers of Alzheimers Disease by Anesthetic Agent Group
Description: CSF Markers of Alzheimer's Disease over time in the subjects treated with propofol versus those treated with isoflurane.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Total Intravenous Anesthesia With Propofol | General Anesthesia With Isoflurane
Number analyzed (Participants) | 55 | 55
pg/ml
  Tau | -0.80 [-26 to 25] | -1.67 [-25 to 32]
  Abeta | -2.10 [-189 to 211] | -9.50 [-127 to 158]
  P-Tau | -2.25 [-31 to 49] | 1.10 [-25 to 85]
Statistical Analysis 1: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Difference in 6-week Tau Change between anesthetic groups; Test type: Other; p = 0.532, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Difference in 6-week Abeta Change between anesthetic groups; Test type: Other; p = 0.565, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Difference in 6-week P-Tau Change between anesthetic groups; Test type: Other; p = 0.110, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Ratio of CSF Markers of Alzheimers Disease by Anesthetic Agent Group
Description: Change in ratio of CSF Markers of Alzheimer's Disease over time in the subjects treated with propofol versus those treated with isoflurane.
Time Frame: baseline to 6-weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: ratio
Arm/Group | Total Intravenous Anesthesia With Propofol | General Anesthesia With Isoflurane
Number analyzed (Participants) | 55 | 55
ratio
  Tau/Abeta Ratio | 0.00 [-0.11 to 0.21] | -0.00 [-0.20 to 0.13]
  P-Tau/Abeta Ratio | -0.00 [-0.10 to 0.28] | 0.01 [-0.08 to 0.41]
Statistical Analysis 1: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Difference in 6-week Tau/Abeta ratio Change between anesthetic groups; Test type: Other; p = 0.439, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Total Intravenous Anesthesia With Propofol vs General Anesthesia With Isoflurane; Difference in 6-week P-Tau/Abeta Change between anesthetic groups; Test type: Other; p = 0.082, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Perioperative CSF Tau/Abeta Ratio Change
Description: The perioperative change in the CSF tau/Abeta ratio from the start of anesthesia/surgery to 24 hours later.
Time Frame: Baseline to 24 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: ratio
Arm/Group | Combined Surgical Cohort
Number analyzed (Participants) | 110
ratio | -0.001 [-0.19 to 0.22]
Statistical Analysis 1: Comparison: Combined Surgical Cohort; Test type: Other; p = 0.801, Wilcoxon Signed Rank

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Non-Surgical Controls: Cohort of community dwelling healthy controls for comparison
Arm/Group | General Anesthesia With Isoflurane | Total Intravenous Anesthesia With Propofol | Non-Surgical Controls
All-Cause Mortality (participants affected / at risk) | 0/72 | 2/68 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/68 | 0/51
Other Adverse Events (participants affected / at risk) | 2/72 | 8/68 | 7/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Anesthesia With Isoflurane (N=72) | Total Intravenous Anesthesia With Propofol (N=68) | Non-Surgical Controls (N=51)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vagal Event (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Leg Pain and Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Post-dural puncture headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Back Pain (General disorders) | 0 (0) | 1 (1) | 3 (5)
Elevated PTT (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Stiffness (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT01993836/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT01993836/SAP_002.pdf